CLINICAL TRIAL: NCT02301806
Title: A Randomized, Prospective, Parallel Design Study to Compare the Effectiveness of Sitagliptin Versus Glimepiride on Endothelial Dysfunction During an Oral Glucose Loading in Drug Naive Patients With Type 2 Diabetes.
Brief Title: Effects of Sitaglpitin on Endothelial Function During the OGTT in T2DM
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Dokkyo Medical University (Other)
Collaborators: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Principal Investigator, Yoshimasa Aso, Professor of Medicine, Dokkyo Medical University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: C-282-02
Record Dates: First submitted 2014-11-22; First posted 2014-11-26 (Estimated); Last update posted 2016-02-17 (Estimated); Status verified 2016-02

CONDITIONS: Type 2 Diabetes
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Sitagliptin Phosphate; glimepiride

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Sitagliptin (Experimental): sitagliptin 50 mg tablet by mouth 12 weeks
  Interventions: Other: dieting; Drug: Sitagliptin
- Glimepiride (Active Comparator): glimepiride 1 mg tablet by mouth 12 weeks
  Interventions: Other: dieting; Drug: Glimepiride

INTERVENTIONS:
Other: dieting
Drug: Sitagliptin — sitagliptin 50 mg tablet by mouth 12 weeks
  Arms: Sitagliptin
Drug: Glimepiride — glimepiride 1 mg tablet by mouth 12 weeks
  Arms: Glimepiride

SUMMARY:
To investigate whether single administration of sitaglitpin can restore acute endothelial dysfunction and ameliorate impaired increase of the number of endothelial progenitor cells (EPCs) after oral glucose loading in patients with T2DM.

To compare the effect of sitagliptin and glimepiride on endothelial function evaluated by flow-mediated vasodilatation (FMD) and the number of circulating EPCs in patients with T2DM.

DETAILED DESCRIPTION:
Acute and chronic improvement of endothelial function is expected through the pleiotropic effect of DPP-4 inhibitors. A randomized, prospective, open-labeled, parallel design. The duration of treatments with sitagliptin or glimepiride is 12 weeks. The number of study centers is a single (Dokkyo Medical University Hospital). Participants will be randomized into the two treatment groups; (a) 50mg sitagliptin (N=15) and (b) 1mg glimepiride (N=15).

Anti-Hyperglycemic effect is expected to be similar according to our study

ELIGIBILITY:
Inclusion Criteria:

* Provision of informed consent before any study specific procedures
* Type II diabetes who have inadequate glycaemic control (6.5%≦HbA1c<9.0%)
* Age from 20 to 80 years old
* No history of using any antihyperglycemic drugs
* No history of cardiovascular complications
* No treatment or treatment with stable doses of lipid-lowering, antihypertensive, and antiplatelet agents for at least 3 months prior to randomization
* 4.5 % ≤ fasting FMD at baseline < 8.0 %

Exclusion Criteria:

* ・Type I diabetes

  * Pregnancy
  * Liver disease (hepatic enzymes more than three times the upper limit of normal ranges)
  * Impairared kidney function (serum crearinine greater than 1.3 mg/dl in men, 1.2 mg/dl in women)
  * Cigarette smokers
  * Contraindications to glimepiride and sitagliptin
  * Active proliferative diabetic retinopathy

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2015-01; Primary Completion 2017-06 (Estimated); Study Completion 2017-07 (Estimated)

PRIMARY OUTCOMES:
Change in endothelial function during the OGTT evaluated by flow-mediated vasodilatation (FMD). The change is defined as below, assuming the peak value and changes of FMD will be observed at t=60 min. | 12 weeks

SECONDARY OUTCOMES:
Change in endothelial function during OGTT* evaluated by endo-PAT. Change in endothelial function after 12-week treatment at the fasting state evaluated by endo-PAT and FMD. | 12 weeks

OTHER OUTCOMES:
Change in the number of EPCs after 12-week treatment | 12 weeeks

CONTACTS AND LOCATIONS:
Overall Officials: Yoshimasa Aso, Principal Investigator — Dokkyo Medical University
Locations (2):
- Japan (2):
  - Dokkyo Medical University, Mibu, Tochigo
  - Mibu